CLINICAL TRIAL: NCT03752034
Title: Safety of Autologous Muscle Fiber Fragments for Improved Function of Rotator Cuff Musculature Following Rotator Cuff Repair
Brief Title: Muscle Fiber Fragments for Improved Function of Rotator Cuff Musculature Following Rotator Cuff Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054333
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Rotator Cuff
Keywords: Muscle Fiber Fragments; Rotator Cuff Musculature; Rotator Cuff Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle Fiber Fragments (MFF) (Experimental): Participants undergoing rotator cuff repair will have autologous muscle tissue harvested. The tissue will be processed to obtain Muscle Fiber Fragments (MFFs) and administered via direct injection into the supraspinatus muscle belly.
  Interventions: Other: Muscle Fiber Fragments (MFFs)

INTERVENTIONS:
Other: Muscle Fiber Fragments (MFFs) — During the rotator cuff repair procedure, a biopsy of muscle will be taken from the pectoralis major and processed under sterile conditions in the operating room to obtain MFFs. The final product, composed of autologous MFFs in suspension, will be delivered via targeted injection into the muscle belly of the supraspinatus through the Naviaser Portal with visual guidance after rotator cuff repair is complete.
  Other Names: Autologous

SUMMARY:
In this study, a chest muscle sample (biopsy) will be taken and the muscle fibers will be removed from the sample and made into smaller strands or fragments. During this same procedure, those muscle fiber fragments (MFFs) will then be injected directly into the supraspinatus muscle. Once injected, the MFFs will remain in the supraspinatus where Investigators believe the MFF will become part of the participants' existing muscle and provide increased muscle size and strength, improving function (rotator cuff strength and stability).

DETAILED DESCRIPTION:
Muscle fiber fragment (MFF) therapy has shown pre-clinical and clinical promise in the treatment of bladder neck insufficiency/incompetent outlet. Fragmentation of muscle fibers derived from autologous muscle tissue can be injected through a needle into the sphincter region. The injected muscle fibers are able to assemble into long muscle fibers in the direction of host muscle fibers. More importantly, muscle progenitor cells residing on the fragmented muscle fibers survive and integrate into host vasculature and nerve to restore damaged muscle function. Preclinical results indicate that this technology can be used to repair and restore damaged sphincter function in urinary incontinence. The development of an autologous, readily available muscle fiber fragment treatment that may involve less risk and recovery time than those associated with the standard surgical therapies and urethral bulking agents, could alter the treatment paradigm of urinary incontinence. The study team hypothesizes that injected MFFs will incorporate into skeletal muscle and re-assemble along the fiber direction. The Investigators anticipate that the MFFs can safely be injected into the atrophied rotator cuff muscle and will help restore the functional contractile properties of the supraspinatus muscle following rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 40 to 80 years
* Unilateral Disease
* < 1.5cm tear

Exclusion Criteria:

* Diabetes
* Peripheral Neuropathy
* Previous Shoulder Surgery
* Pain Syndrome; cuff arthroplasty
* Major co-morbidities including, but not limited to, uncontrolled diabetes, cardiovascular, pulmonary, GI, coagulopathies
* Arthritis of Shoulder
* Unwilling or unable to comply with post-operative instructions or follow-up visits
* Auto Immune Disease
* Complete Subscapularis Tear
* Teres Minor involvement
* History of testing positive for HIV, Hep B, Hep C, HTLV-1, HTLV-2
* Pregnancy
* Implanted devices containing ferromagnetic material
* Any implanted electrical stimulation devices (i.e. cochlear implant, defibrillator)
* Any other condition which the PI feels would be not in the best interest for the patient or the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 6 months post surgery
  The incidence of adverse events will be documented in the areas of product related, biopsy procedure-related, and injection-related reporting for each group.
Incidence of Adverse Events | 12 months post surgery
  The incidence of adverse events will be documented in the areas of product related, biopsy procedure-related, and injection-related reporting for each group.

SECONDARY OUTCOMES:
Fat Free Muscle Volume | Month 1, Month 6, and Month 12
  Fat-free muscle volume (total muscle volume minus % of fatty infiltration).
Goutallier Score via MRI 1.5+ image analysis | 12 weeks, 6 months, and 12 months post operatively
  Measured by MRI T1 Sagittal image at the Y position. Total score values 0- 4 (Grade 0 =normal muscle; Grade 1 =Muscle that contain some fatty streaks; Grade 2 = Fatty infiltration but more muscle than fat; Grade 3 = Equal amounts of fat and muscle; Grade 4 = More fat than muscle.) Lower values denotes better outcomes.
Constant Score | 12 weeks, 6 months, and 12 months post operatively
  The constant score, a 0-100 point scale with 100 being Normal and Abnormal Side >30 Poor, 21-30 Fair, 11-20 Good and <11 Excellent will measure muscle recovery including strength and level of atrophy. Higher scores denote worse outcome measures.
ASES Shoulder Score | 12 weeks, 6 months, and 12 months post operatively
  The ASES Shoulder Score (scale with a max of 100 which is normal function with no pain to minimum of 0 which is extreme pain) will measure muscle recovery. Higher scores denote better outcomes.
Dynamometer measurements | 12 weeks, 6 months, and 12 months post operatively
  Measurement will be on a scale used to measure the number of pounds or kilograms generated with arm at 90 degrees of abduction with the elbow extended.

CONTACTS AND LOCATIONS:
Overall Officials: Gary G Poehling, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deniz G, Kose O, Tugay A, Guler F, Turan A. Fatty degeneration and atrophy of the rotator cuff muscles after arthroscopic repair: does it improve, halt or deteriorate? Arch Orthop Trauma Surg. 2014 Jul;134(7):985-90. doi: 10.1007/s00402-014-2009-5. Epub 2014 May 21. PMID 24845686
- [Background] Eberli D, Aboushwareb T, Soker S, Yoo JJ, Atala A. Muscle precursor cells for the restoration of irreversibly damaged sphincter function. Cell Transplant. 2012;21(9):2089-98. doi: 10.3727/096368911X623835. Epub 2012 Jan 10. PMID 22236637
- [Background] Eberli D, Andersson KE, Yoo JJ, Atala A. A canine model of irreversible urethral sphincter insufficiency. BJU Int. 2009 Jan;103(2):248-53. doi: 10.1111/j.1464-410X.2008.08001.x. Epub 2008 Sep 8. PMID 18782310
- [Background] MAURO A. Satellite cell of skeletal muscle fibers. J Biophys Biochem Cytol. 1961 Feb;9(2):493-5. doi: 10.1083/jcb.9.2.493. No abstract available. PMID 13768451
- [Background] Benchaouir R, Rameau P, Decraene C, Dreyfus P, Israeli D, Pietu G, Danos O, Garcia L. Evidence for a resident subset of cells with SP phenotype in the C2C12 myogenic line: a tool to explore muscle stem cell biology. Exp Cell Res. 2004 Mar 10;294(1):254-68. doi: 10.1016/j.yexcr.2003.11.005. PMID 14980519
- [Background] Partridge TA, Morgan JE, Coulton GR, Hoffman EP, Kunkel LM. Conversion of mdx myofibres from dystrophin-negative to -positive by injection of normal myoblasts. Nature. 1989 Jan 12;337(6203):176-9. doi: 10.1038/337176a0. PMID 2643055
- [Background] Yiou R, Lefaucheur JP, Atala A. The regeneration process of the striated urethral sphincter involves activation of intrinsic satellite cells. Anat Embryol (Berl). 2003 May;206(6):429-35. doi: 10.1007/s00429-003-0313-x. Epub 2003 May 1. PMID 12728313
- [Background] Gussoni E, Soneoka Y, Strickland CD, Buzney EA, Khan MK, Flint AF, Kunkel LM, Mulligan RC. Dystrophin expression in the mdx mouse restored by stem cell transplantation. Nature. 1999 Sep 23;401(6751):390-4. doi: 10.1038/43919. PMID 10517639
- [Background] Leobon B, Garcin I, Menasche P, Vilquin JT, Audinat E, Charpak S. Myoblasts transplanted into rat infarcted myocardium are functionally isolated from their host. Proc Natl Acad Sci U S A. 2003 Jun 24;100(13):7808-11. doi: 10.1073/pnas.1232447100. Epub 2003 Jun 12. PMID 12805561
- [Background] Seidel M, Borczynska A, Rozwadowska N, Kurpisz M. Cell-based therapy for heart failure: skeletal myoblasts. Cell Transplant. 2009;18(7):695-707. doi: 10.3727/096368909X470810. Epub 2009 Apr 6. PMID 19500482
- [Background] Yiou R, Yoo JJ, Atala A. Restoration of functional motor units in a rat model of sphincter injury by muscle precursor cell autografts. Transplantation. 2003 Oct 15;76(7):1053-60. doi: 10.1097/01.TP.0000090396.71097.C2. PMID 14557752
- [Background] Badra S, Andersson KE, Dean A, Mourad S, Williams JK. Long-term structural and functional effects of autologous muscle precursor cell therapy in a nonhuman primate model of urinary sphincter deficiency. J Urol. 2013 Nov;190(5):1938-45. doi: 10.1016/j.juro.2013.04.052. Epub 2013 Apr 22. PMID 23618586